CLINICAL TRIAL: NCT03035916
Title: Effect of Transversus Abdominis Plane Block Combined With General Anesthesia on Perioperative Stress Response in Patients Undergoing Radical Gastrectomy: A Double-blind Randomized Controlled Study.
Brief Title: Transversus Abdominis Plane Block on Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Zhao Guoqing, Clinical Professor, Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3D5l4L463430; 3R210Z893430 (Other Grant/Funding Number: Jilin Provincial Department of Science and Technology)
Record Dates: First submitted 2017-01-13; First posted 2017-01-30 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Gastrostomy
Keywords: transversus abdominal plane block; epidural anesthesia; stress response; anesthetic recovery
MeSH Terms: conditions — Fractures, Stress | interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus abdominis plane block (Experimental): The TAP group receives ultrasound-guided TAP block under bilateral costal margin with multiple injections of 40ml 0.375% ropivacaine after the induction of general anesthesia.
  Interventions: Other: Transversus abdominis plane block
- Epidural anesthesia (Active Comparator): The Epidural group receives epidural block (T8-9) 2 mL of 1.6% lidocaine as a test dose and continous infusion of 0.375% ropivacaine(5 mL/h) during the surgery.
  Interventions: Other: Epidural anesthesia
- Control (Placebo Comparator): The Control group receives standard IV-inhaled general anesthesia.
  Interventions: Other: control

INTERVENTIONS:
Other: Transversus abdominis plane block — Participants in this group receive ultrasound-guided TAP block under bilateral costal margin with multiple injections of 40ml 0.375% ropivacaine after the induction of general anesthesia, 30 minutes later the surgery will be started.
  Arms: Transversus abdominis plane block
Other: Epidural anesthesia — Participants in the Epidural group receive a epidural block (T8-9) with 2 mL of 1.6% lidocaine as a test dose before induction. After a successful placement of epidural catheter, the block then is established with 5 mL of 0.375% ropivacaine and continous infusion of 0.375% ropivacaine(5 mL/h) during the surgery.
  Arms: Epidural anesthesia
Other: control — The Control group receives standard IV-inhaled general anesthesia.
  Arms: Control

SUMMARY:
This study evaluates the effect of transversus abdominis plane(TAP) block combined with general anesthesia on perioperative stress response in patients undergoing radical gastrectomy. One third of participants will receive TAP block combined with general anesthesia, another one third of participants will receive epidural anesthesia combined with general anesthesia, while the rest will receive only general anesthesia.

DETAILED DESCRIPTION:
Clinically, combining epidural with general anaesthesia may confer many advantages to patients undergoing major thoracic, abdominal or orthopaedic surgery. Epidural anaesthesia can attenuate sympathetic hyperactivity and the stress response, maintain bowel peristalsis, spare the use of opioids, and facilitate postoperative feeding and physiotherapy. However, establishing epidural anesthesia is not without risks and contraindications, including refusal by the patient, technical failure, unintentional dural puncture, waist and back pain and local anaesthetic toxicity. When neurologic complications do occur, the resulting morbidity and mortality is considerable. Transversus abdominis plane (TAP) block, is another new regional anesthesia technique, has been introduced as an abdominal wall block capable of providing effective analgesia, reducing opioid consumption, and lessening opioid-related side effects. In addition,TAP block, somewhat as a pre-emptive analgesia approach, is a way of pain intervention before noxious stimulation which has been reported to be potent to attenuate the stress response. Although the analgesia efficiency of TAP block has been widely studied, its effectiveness to suppress stress response has little comparison with classic epidural block and general anesthesia. Unlike epidural anaesthesia, TAP block is easy to administer and lower incidence for side-effects.The investigators hypothesize that the TAP block reduces the stress response of surgery to the similar extent to epidural anaesthesia when combined with a standard general anaesthesia for abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* ASA 1-3
* No contraindication to epidural or ropivacaine
* First time surgery for current conditions
* Not on chronic pain medications or sedative

Exclusion Criteria:

* The subject has a known or suspected allergy to opioid analgesics or ropivacaine
* Emergency patients
* The subject has know central nervous system disease or neurological impairment
* The subject has preoperative infection, and a history of immune and endocrine system disease, chemotherapy, or blood transfusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Zhao, doctor, Principal Investigator — Jilin University
Locations (1):
- China-Japan Union Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to the analysis by PASS 11.0, at lease 25 participants each arm were needed.Taking into account the withdrawal of patients in the middle of the study, each group were more than a few included
Period: Overall Study
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Started | 30 | 30 | 31
Completed | 30 | 28 | 31
Not Completed | 0 | 2 | 0
Not completed — Puncture failed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control | Total
Number analyzed (Participants) | 30 | 28 | 31 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 21 | 63
  >=65 years | 8 | 8 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.75 (8.24) | 58.60 (8.72) | 60.20 (9.43) | 59.18 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 25
  Male | 21 | 20 | 23 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 30 | 28 | 31 | 89
ASA physical status [Count of Participants; unit: Participants] — ASA I: No organic, physiologic, biochemical or psychiatric disturbance; ASA II: A patient with mild systemic disease that results in no functional limitation; ASA III: A patient with severe systemic disease that results in functional impairment; ASA IV: Severe systemic disease that is a constant threat to life; ASA V: Moribund condition in a patient who is not expected to survive with or without the operation; ASA VI: Declared brain death patient whose organs are being harvested for transplantation; E: Emergency operation is required.
  Participants
    I | 5 | 4 | 4 | 13
    II | 19 | 18 | 20 | 57
    III | 6 | 6 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Physiological Parameters: Plasma Concentration of Norepinephrine (NE)
Description: Venous blood samples will be collected at certain time points. The blood samples are collected in a pre-chilled tubes in ice and are centrifuged within 90min, and then separated plasma are stored at -80°C until analysis. The NE levels are measured by ELISA kits.
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
pg/ml
  Baseline | 145.6 (25.8) | 150.9 (33.2) | 153.1 (35.2)
  0 hr after surgery | 170.2 (33.4) | 165.5 (36.6) | 177.9 (43.2)
  6 hr after surgery | 172.3 (32.7) | 163.2 (32.4) | 215.5 (50.3)
  24 hr after surgery | 150.5 (30.9) | 155.8 (25.3) | 175.4 (40.2)
  48 hr after surgery | 135.7 (29.8) | 140.6 (24.8) | 165.2 (32.7)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of norepinephrine(NE) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.454, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.402, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.901, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of norepinephrine(NE) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "0 hour after surgery" row; Test type: Other; p = 0.540, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.523, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.260, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of norepinephrine(NE) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.139, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 1, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 1, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of norepinephrine(NE) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.464, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 1, analysis 10]; Test type: Other; p = 0.007, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 1, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of norepinephrine(NE) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.411, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 1, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 1, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided

2. Primary Outcome: Physiological Parameters: Plasma Concentration of Epinephrine (E)
Description: Venous blood samples will be collected at certain time points. The blood samples are collected in a pre-chilled tubes in ice and are centrifuged within 90min, and then separated plasma are stored at -80°C until analysis. The E levels are measured by ELISA kits.
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
pg/ml
  Baseline | 33.2 (6) | 35 (5.4) | 34.4 (6.1)
  0 hr after surgery | 41.5 (6.6) | 40.5 (7.2) | 42.2 (7)
  6 hr after surgery | 45.3 (8.2) | 46.4 (7.5) | 52.3 (8.1)
  24 hr after surgery | 44.5 (7) | 41.8 (6.2) | 59.1 (8.5)
  48 hr after surgery | 40.6 (6.3) | 39.3 (5.2) | 48.7 (7.6)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of epinephrine (E) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.412, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.592, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.796, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of epinephrine (E) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "0 hour after surgery" row; Test type: Other; p = 0.576, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.427, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = 0.201, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of epinephrine (E) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.872, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 2, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 2, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of epinephrine (E) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.165, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 2, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 2, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of epinephrine (E) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control. This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.305, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 2, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 2, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided

3. Primary Outcome: Physiological Parameters: Plasma Concentration of Cortisol (Cor)
Description: Venous blood samples will be collected at certain time points. The blood samples are collected in a pre-chilled tubes in ice and are centrifuged within 90min, and then separated plasma are stored at -80°C until analysis. The Cor levels are measured by ELISA kits.
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
mmol/L
  Baseline | 273.3 (93) | 262.4 (101.5) | 286.3 (106.6)
  0 hr after surgery | 430.4 (152.1) | 395.2 (133.4) | 516.1 (162.3)
  6 hr after surgery | 519.2 (156.6) | 464.2 (155.8) | 698.3 (188.1)
  24 hr after surgery | 439 (116) | 388.1 (121.2) | 713.8 (190)
  48 hr after surgery | 320.6 (112.3) | 302.8 (112.4) | 452.4 (165.3)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of cortisol (Cor) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.673, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.824, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.547, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of cortisol (Cor) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "0 hour after surgery" row; Test type: Other; p = 0.303, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 3, analysis 4]; Test type: Other; p = 0.026, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 3, analysis 4]; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of cortisol (Cor) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.057, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 3, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 3, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of cortisol (Cor) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.069, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 3, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 3, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of cortisol (Cor) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.561, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 3, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 3, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided

4. Primary Outcome: Physiological Parameters: Plasma Concentration of Glucose (Glu)
Description: When venous blood are collected, glucose levels are measured immediately by Glucometer.
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
mmol/L
  Baseline | 5 (0.5) | 5.2 (0.5) | 5.5 (0.4)
  0 hr after surgery | 8.2 (1.2) | 7.7 (0.9) | 10.5 (1.5)
  6 hr after surgery | 7.5 (1) | 7 (0.9) | 10.8 (1.9)
  24 hr after surgery | 6.5 (0.8) | 6.3 (0.7) | 8.6 (1.5)
  48 hr after surgery | 5.5 (0.4) | 5.2 (0.5) | 5.8 (0.6)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.249, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.091, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.493, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "0 hour after surgery" row; Test type: Other; p = 0.067, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 4, analysis 4]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 4, analysis 4]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.079, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 4, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 4, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.314, t-test, 2 sided — The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "24 hours after surgery" row
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 4, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 4, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The plasma level of glucose (Glu) were detected from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.087, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 4, analysis 13]; Test type: Other; p = 0.023, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 4, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided

5. Primary Outcome: Hemodynamic Parameters: Heart Rate.
Description: Continuous monitoring of heart rate to 48 hours after surgery.
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
bpm
  Baseline | 75.4 (12.5) | 77.1 (11.1) | 76.4 (12)
  Before induction | 74.8 (10.9) | 70 (12.2) | 76 (11)
  Induction | 71.1 (10.8) | 63.1 (10.3) | 71.7 (10.2)
  Intubation | 88.4 (11.5) | 87 (13) | 92 (13.5)
  Incision | 80 (11.4) | 78 (11.5) | 95.7 (13.3)
  Extubation | 82 (13.5) | 80 (13) | 85 (15)
  6 hr after surgery | 77 (10.5) | 75 (10) | 79 (12)
  24 hr after surgery | 75 (10.9) | 74 (11) | 81.3 (10.8)
  48 hr after surgery | 75.8 (10.3) | 75 (10.5) | 79.5 (11.5)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.384, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.530, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.819, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Before induction" row; Test type: Other; p = 0.108, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 4]; Test type: Other; p = 0.667, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 4]; Test type: Other; p = 0.046, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Induction" row; Test type: Other; p = 0.006, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 7]; Test type: Other; p = 0.406, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 7]; Test type: Other; p = 0.042, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Intubation" row; Test type: Other; p = 0.655, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 10]; Test type: Other; p = 0.262, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 10]; Test type: Other; p = 0.143, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Incision" row; Test type: Other; p = 0.494, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 16: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Extubation" row; Test type: Other; p = 0.555, t-test, 2 sided
Statistical Analysis 17: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 16]; Test type: Other; p = 0.411, t-test, 2 sided
Statistical Analysis 18: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 16]; Test type: Other; p = 0.167, t-test, 2 sided
Statistical Analysis 19: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.445, t-test, 2 sided
Statistical Analysis 20: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 19]; Test type: Other; p = 0.489, t-test, 2 sided
Statistical Analysis 21: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 19]; Test type: Other; p = 0.159, t-test, 2 sided
Statistical Analysis 22: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.720, t-test, 2 sided
Statistical Analysis 23: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 22]; Test type: Other; p = 0.026, t-test, 2 sided
Statistical Analysis 24: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 22]; Test type: Other; p = 0.011, t-test, 2 sided
Statistical Analysis 25: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The Heart rate was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.763, t-test, 2 sided
Statistical Analysis 26: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 5, analysis 25]; Test type: Other; p = 0.187, t-test, 2 sided
Statistical Analysis 27: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 5, analysis 25]; Test type: Other; p = 0.112, t-test, 2 sided

6. Primary Outcome: Hemodynamic Parameters: Mean Arterial Pressure(MAP)
Description: Continuous monitoring of mean arterial pressure(MAP) to 48 hours after surgery. mean arterial pressure(MAP)＝ (systolic blood pressure＋2×diastolic blood pressure)/3
Time Frame: up to 48h after surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
mmHg
  Baseline | 87 (12.5) | 88.5 (11) | 86 (12)
  Before induction | 90 (13) | 80 (12) | 87 (13)
  Induction | 81 (10.5) | 73 (12) | 80 (13)
  Intubation | 93 (13.5) | 90 (15) | 94 (15.5)
  Incision | 85 (12) | 84 (11.5) | 98 (15)
  Extubation | 88 (13.5) | 90 (13) | 95 (15)
  6 hr after surgery | 89 (10.5) | 86 (10) | 93 (12)
  24 hr after surgery | 88 (12.5) | 84 (11) | 90 (14)
  48 hr after surgery | 89 (12) | 85 (10.5) | 90 (11.5)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Baseline" row; Test type: Other; p = 0.645, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.645, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.314, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Before induction" row; Test type: Other; p = 0.003, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 4]; Test type: Other; p = 0.367, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 4]; Test type: Other; p = 0.031, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Induction" row; Test type: Other; p = 0.009, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 7]; Test type: Other; p = 0.873, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 7]; Test type: Other; p = 0.026, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Intubation" row; Test type: Other; p = 0.411, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 10]; Test type: Other; p = 0.787, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 10]; Test type: Other; p = 0.306, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Incision" row; Test type: Other; p = 0.921, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 16: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "Extubation" row; Test type: Other; p = 0.555, t-test, 2 sided
Statistical Analysis 17: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 16]; Test type: Other; p = 0.058, t-test, 2 sided
Statistical Analysis 18: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 16]; Test type: Other; p = 0.166, t-test, 2 sided
Statistical Analysis 19: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.288, t-test, 2 sided
Statistical Analysis 20: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 19]; Test type: Other; p = 0.299, t-test, 2 sided
Statistical Analysis 21: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 19]; Test type: Other; p = 0.051, t-test, 2 sided
Statistical Analysis 22: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.186, t-test, 2 sided
Statistical Analysis 23: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 22]; Test type: Other; p = 0.555, t-test, 2 sided
Statistical Analysis 24: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 22]; Test type: Other; p = 0.065, t-test, 2 sided
Statistical Analysis 25: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The mean arterial pressure(MAP) was measured from baseline to 48hours after surgery. The row "Baseline" is the preoperative level as the blank control.This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.168, t-test, 2 sided
Statistical Analysis 26: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 6, analysis 25]; Test type: Other; p = 0.739, t-test, 2 sided
Statistical Analysis 27: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 6, analysis 25]; Test type: Other; p = 0.079, t-test, 2 sided

7. Secondary Outcome: Anesthetics Consumption: Sufentanil Consumption
Description: Intraoperative superaddition of sufentanil was measured.
Time Frame: during operation
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
ug | 4.3 (1.5) | 3.6 (1.2) | 10.2 (2.8)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.056, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.001, t-test, 2 sided

8. Secondary Outcome: Questionnaire: Pain Scores at Rest
Description: Pain scores of the participants will be measured by the Visual Analogue Scale. Measurement of VAS: Draw a 10cm horizontal line on the paper. The VAS were anchored at 0cm(no pain) and 10cm(worst possible pain), the middle part shows varying degrees of pain, the greater of the number, the worse of the pain.
Time Frame: 1hr, 6hr, 12hr, 24hr, and 48hr after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
units on a scale
  1 hr | 2.2 (0.7) | 1.8 (1.0) | 2.7 (0.6)
  6 hr | 2.2 (0.9) | 1.9 (0.8) | 2.7 (1.0)
  12 hr | 2.0 (0.7) | 1.7 (0.7) | 2.8 (1.0)
  24 hr | 2.2 (0.6) | 1.3 (0.6) | 2.7 (1.0)
  48 hr | 1.0 (0.8) | 0.9 (0.6) | 1.3 (0.8)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The pain score were measured from 1 hour to 48hours after surgery. This Statistical Analysis applied to "1 hour after surgery" row; Test type: Other; p = 0.056, t-test, 2 sided — p<0.05 indicates that the data difference is statistically significant
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.009, t-test, 2 sided — p<0.05 indicates that the data difference is statistically significant
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.001, t-test, 2 sided — p<0.05 indicates that the data difference is statistically significant
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The pain score were measured from 1 hour to 48hours after surgery. This Statistical Analysis applied to "6 hours after surgery" row; Test type: Other; p = 0.198, t-test, 2 sided
Statistical Analysis 5: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 4]; Test type: Other; p = 0.047, t-test, 2 sided
Statistical Analysis 6: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 4]; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The pain score were measured from 1 hour to 48hours after surgery. This Statistical Analysis applied to "12 hours after surgery" row; Test type: Other; p = 0.102, t-test, 2 sided
Statistical Analysis 8: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.005, t-test, 2 sided
Statistical Analysis 9: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The pain score were measured from 1 hour to 48hours after surgery. This Statistical Analysis applied to "24 hours after surgery" row; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 11: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 10]; Test type: Other; p = 0.023, t-test, 2 sided
Statistical Analysis 12: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; The pain score were measured from 1 hour to 48hours after surgery. This Statistical Analysis applied to "48 hours after surgery" row; Test type: Other; p = 0.425, t-test, 2 sided
Statistical Analysis 14: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 13]; Test type: Other; p = 0.124, t-test, 2 sided
Statistical Analysis 15: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 13]; Test type: Other; p = 0.052, t-test, 2 sided

9. Secondary Outcome: Questionnaire: Pain Scores on Movement
Description: as for outcome 8
Time Frame: 1hr, 6hr, 12hr, 24hr, and 48hr after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
units on a scale
  1 hr | 2.7 (1.2) | 2.4 (1.1) | 4.3 (0.8)
  6 hr | 2.9 (0.7) | 2.6 (1.3) | 4.2 (0.7)
  12 hr | 3.3 (0.5) | 3.7 (0.9) | 4.0 (0.8)
  24 hr | 4.1 (0.7) | 3.5 (0.9) | 4.6 (0.8)
  48 hr | 4.2 (0.8) | 3.5 (0.8) | 4.5 (0.9)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.176, t-test, 2 sided — p<0.05 indicates that the data difference is statistically significant
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.001, t-test, 2 sided — p<0.05 indicates that the data difference is statistically significant
Statistical Analysis 3: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; [analysis description as in outcome 8, analysis 4]; Test type: Other; p = 0.228, t-test, 2 sided
Statistical Analysis 4: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 4]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 4]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 6: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.057, t-test, 2 sided
Statistical Analysis 7: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 8: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 9: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; [analysis description as in outcome 8, analysis 10]; Test type: Other; p = 0.004, t-test, 2 sided
Statistical Analysis 10: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 10]; Test type: Other; p = 0.005, t-test, 2 sided
Statistical Analysis 11: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 10]; Test type: Other; p = 0.001, t-test, 2 sided
Statistical Analysis 12: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; [analysis description as in outcome 8, analysis 13]; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 13: Comparison: Transversus Abdominis Plane Block vs Control; [analysis description as in outcome 8, analysis 13]; Test type: Other; p = 0.002, t-test, 2 sided
Statistical Analysis 14: Comparison: Epidural Anesthesia vs Control; [analysis description as in outcome 8, analysis 13]; Test type: Other; p = 0.001, t-test, 2 sided

10. Secondary Outcome: Anesthesia Recovery: the Time of First Flatus
Description: The time of first flatus was measured after surgery.
Time Frame: Through study completion, an average of 2 weeks
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
hour | 77.6 (10.4) | 78.4 (11.6) | 81.6 (10.4)
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.585, t-test, 2 sided
Statistical Analysis 2: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.071, t-test, 2 sided
Statistical Analysis 3: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.13, t-test, 2 sided

11. Secondary Outcome: Anesthesia Recovery: Number of Participants With Prolonged Hospitalization
Description: The percentage of long hospitalization were measured. More than 7 days after surgery is defined as prolonged hospitalization.
Time Frame: Through study completion, an average of 2 weeks
Measure: Number; unit: participants
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
participants | 5 | 5 | 13
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.644, t-test, 2 sided
Statistical Analysis 2: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.045, t-test, 2 sided
Statistical Analysis 3: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.031, t-test, 2 sided

12. Secondary Outcome: Side Effects: Number of Participants With Sedation
Description: The state of sedation was evaluated after surgery during first postoperative 48 hours.
Time Frame: up to 48h after surgery
Measure: Number; unit: participants
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
participants | 8 | 5 | 16
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.421, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.046, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.007, t-test, 2 sided

13. Secondary Outcome: Side Effects: Number of Participants With Nausea
Description: The state of nausea was evaluated after surgery during first postoperative 48 hours.
Time Frame: up to 48h after surgery
Measure: Number; unit: participants
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
participants | 5 | 4 | 6
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.910, t-test, 2 sided
Statistical Analysis 2: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.864, t-test, 2 sided
Statistical Analysis 3: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.785, t-test, 2 sided

14. Secondary Outcome: Side Effects: Number of Participants With Vomiting
Description: The state of vomiting was evaluated after surgery during first postoperative 48 hours.
Time Frame: up to 48h after surgery
Measure: Number; unit: participants
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
Number analyzed (Participants) | 30 | 28 | 31
participants | 0 | 1 | 1
Statistical Analysis 1: Comparison: Transversus Abdominis Plane Block vs Epidural Anesthesia; Test type: Other; p = 0.972, t-test, 2 sided
Statistical Analysis 2: Comparison: Transversus Abdominis Plane Block vs Control; Test type: Other; p = 0.987, t-test, 2 sided
Statistical Analysis 3: Comparison: Epidural Anesthesia vs Control; Test type: Other; p = 0.518, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Transversus Abdominis Plane Block | Epidural Anesthesia | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 2/28 | 0/31
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transversus Abdominis Plane Block (N=30) | Epidural Anesthesia (N=28) | Control (N=31)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Firstly, early termination leading to small numbers of subjects analyzed. Secondly, sufentanil for analgesia, known to have effects on neuroimmunoendocrine network, which may have influenced our finding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03035916/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03035916/SAP_001.pdf
  • Informed Consent Form (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03035916/ICF_002.pdf